CLINICAL TRIAL: NCT04388566
Title: Development of the Danish Prospective Sarcoidosis Registry and Baseline Characteristics of a Danish Sarcoidosis Cohort
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: SAR1
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-09

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Development of a Danish Sarcoidosis Registry. Characterization of a cohort of sarcoidosis patients with respect to the baseline epidemiological characteristics, comorbidities, radiology, histopathology, diagnostic investigations and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis
* Signed informed consent

Exclusion Criteria:

* Inability or unwillingness to adhere to the study
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sarcoidosis seen in the Department of Respiratory Diseases, Aarhus Denmark
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Characterization of Danish sarcoid patients | 2 years
  Epidemiology and Baseline characteristics of a Danish Sarcoidosis Cohort
Feasibility and completion of a Sarcoidosis Registry. | 2 years
  Development of a Danish sarcoidosis registry Data on epidemiology, clinical characteristics, diagnosis and management will be registered

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark